CLINICAL TRIAL: NCT06545253
Title: A New Diagnostic Paradigm for Retinitis Pigmentosa Secondary to USH2A Pathogenic Variants
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Maria Lucia Cascavilla, Co-Principal Investigator, IRCCS Ospedale San Raffaele
Other Study IDs: PNRR-MR1-2023-12378435
Record Dates: First submitted 2024-07-14; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: USH2A Variant Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- USH2A-RP: Patients affected by genetically-confirmed USH2A-RP.
  Interventions: Diagnostic Test: microRNAs analysis
- controls: Healthy control subjects
  Interventions: Diagnostic Test: microRNAs analysis

INTERVENTIONS:
Diagnostic Test: microRNAs analysis — Patients will undergo routinary ophthalmological examination, multimodal retinal imaging and blood sampling
  Other Names: multimodal retinal imaging

SUMMARY:
Aim of the study is to perform a non-invasive multimodal retinal imaging investigation in a cohort of patients affected by USH2A retinitis pigmentosa (USH2A-RP), in order to develop a new diagnostic paradigm to categorize clinically relevant subgroups. All the procedures will be performed according to normal clinical practice. In addition, a novel quantitative profiling of serum microRNAs will be carried out in order to analyze the clinical importance of microRNA biomarkers in the clinical setting of the disease.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* genetically confirmed diagnosis of USH2A-RP
* availability of genetic tests to assess the pathogenic variants

Exclusion Criteria:

* inability to understand and sign the written informed consent form
* any inflammatory, infectious or degenerative eye disease
* media opacities resulting incompatible with good imaging quality
* uncontrolled systemic, metabolic, autoimmune neuroinflammatory and neurodegenerative disease
* ophthalmologic surgery within the previous six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * 60 patients affected by genetically-confirmed USH2A-RP, both males and females, age >18 years
  * 10 healthy age- and gender- matched control subjects recruited among healthy patients undergoing general ophthalmological examinations in the outpatient departments
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Clinical relevance of microRNAs in USH2A-RP | 6 months period following the last follow-up visit
  For all patients enrolled, at baseline, peripheral blood sampling will be collected.

SECONDARY OUTCOMES:
To test the association between specific microRNAs profiles and the quantitative multimodal retinal imaging findings | 6 months period following the last follow-up visit
  At baseline and month 12 follow-up visit, all enrolled patients with a genetically confirmed diagnosis of USH2A-RP, will undergo the following procedures:
  * complete ophthalmic examination, including best corrected visual acuity measurement using standard ETDRS charts, intraocular pressure, slit-lamp biomicroscopy of the anterior and posterior segment;
  * multimodal retinal imaging including: Ultrawide field imaging either with Optos devices; Blue-light fundus autofluorescence (FAF); Infrared imaging (IR); Multicolor imaging with Spectralis SD-OCT; Optical coherence tomography (OCT) with Spectralis SD-OCT; Optical coherence tomography angiography (OCTA) of the macula; visual field with standard 30.2 test pattern by Humphrey field analyzer.